CLINICAL TRIAL: NCT04640714
Title: Care Transition Intervention for Hospitalized Patients With Advanced Cancer
Brief Title: Care Transition Intervention for Patients With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jennifer Temel, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-418
Record Dates: First submitted 2020-11-11; First posted 2020-11-23 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Advanced Cancer; Home Care, Hospital-Based
Keywords: Advanced Cancer; Home Care, Hospital-Based; Transitions of Care; Care Transition Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CONTINUity of care Under Management by Video visits (CONTINUUM-V) (Experimental): Participants with advanced cancer will receive a video visit conducted by an oncology Nurse Practitioner (NP) within three (3) business days of hospital discharge.
  The visit will involve: (1) reconcile medications, (2) manage symptoms, (3) review the post-hospital care plan for hospitalization-specific issues, and (4) schedule follow-up with the outpatient oncology team.
  Participant and clinician may also be interviewed for their feedback on the video visit.
  The ultimate goal of the intervention is to improve patients' confidence in managing their health condition and reduce burdensome health care utilization after discharge, particularly reducing 30-day hospital readmissions.
  Interventions: Behavioral: CONTINUity of care Under Management by Video visits (CONTINUUM-V)

INTERVENTIONS:
Behavioral: CONTINUity of care Under Management by Video visits (CONTINUUM-V) — Video visit by nurse practitioner within 3 business days of hospital discharge.

SUMMARY:
This research study is investigating an intervention called CONTINUity of care Under Management by Video visits (CONTINUUM-V). CONTINUUM-V involves a video visit with an oncology nurse practitioner within three business days of hospital discharge for patients with advanced cancer with the goal of reducing burdensome care transitions after hospitalization, including hospital readmissions.

DETAILED DESCRIPTION:
This is a single-site, single-arm pilot trial to assess the feasibility and acceptability of a CONTINUUM-V for patients with advanced cancer

The research study procedures include:

* A video visit with a nurse practitioner within three business days of hospital discharge
* Questionnaires asking about demographic information (e.g. sex, ethnicity, income) and participant experience with cancer (e.g. symptoms and confidence in managing their health condition)
* A satisfaction survey to assess the participants' impressions of the intervention and any suggestions the participants may have
* Data collection from their medical record
* One time interview of participant and clinician for feedback on CONTINUUM-V

Participants will be in this research study for up to 45 days after hospital discharge.

54 patients and 4 clinicians took part in this research study.

The Conquer Cancer Foundation and the Rising Tide Foundation for Clinical Cancer Research are supporting this research study by providing a Career Pathway Grant in Symptom Management to support the research team.

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 18 years
2. Unplanned admission to the oncology service at Massachusetts General Hospital (MGH)
3. Known diagnosis of advanced breast, thoracic, genitourinary, or gastrointestinal cancers. Advanced cancer defined as not being treated with curative intent as determined by clinic notes and chemotherapy order entry.
4. Receiving ongoing oncology care at MGH
5. Verbal fluency in English
6. Must have internet/wifi/cellular data access

Exclusion Criteria:

1. Admitted electively
2. Discharged to a location other than home or expired during admission
3. Discharged with hospice services

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2021-01-07 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2021-07-14 (Actual)

PRIMARY OUTCOMES:
Feasibility using enrollment and retention on study | Discharge to 3 business days
  The intervention will be deemed feasible if at least 70% of eligible patients participate in the study, and if at least 70% complete the video visit within three business days of discharge.

SECONDARY OUTCOMES:
Patients' Confidence in Managing their Health Condition using the Patient Activation Measure (PAM-13) | Baseline to 15 days after discharge
  The investigators will use the Patient Activation Measure 13 (PAM-13) to assess participants' confidence in managing their health condition at baseline and within 10-15 days of discharge (post-intervention). The PAM-13 is scored 0-100 with higher scores indicating greater confidence in managing one's health condition.
Symptom Burden using the Edmonton Symptom Assessment Scale (ESAS-r) | Baseline to 15 days after discharge
  The investigators will use a modified version of the self-administered, revised Edmonton Symptom Assessment System (ESAS-r) to assess participants' symptoms at baseline and within 10-15 days of discharge (post-intervention). The ESAS-r assesses pain, fatigue, drowsiness, nausea, appetite, dyspnea, depression, anxiety, and well being over the previous 24 hours. The ESAS-r also includes constipation. Individual symptoms are scored on a scale from 0 (reflecting absence of the symptom) to 10 (reflecting the worst possible severity). The investigators will compute the composite ESAS physical and total symptom variables that included scores of participants' physical symptoms (pain, fatigue, drowsiness, nausea, appetite, dyspnea, constipation) and total symptoms (pain, fatigue, drowsiness, nausea, appetite, dyspnea, depression, anxiety, well being, constipation).
Psychological Symptoms using the Patient Health Questionnaire-4 (PHQ-4) | Baseline to 15 days after discharge
  The investigators will use the Patient Health Questionnaire-4 (PHQ-4) to assess psychological symptoms at baseline and within 10-15 days of discharge (post-intervention). The PHQ-4 is a 4-item tool that contains two 2-item subscales assessing depression and anxiety symptoms. Both subscales and the composite PHQ-4 score can also be evaluated continuously, with higher scores indicating worse psychological distress. Scores on each subscale range from 0 to 6.
Patient Satisfaction using the Patient Satisfaction Questionnaire | 10 to 15 days after discharge
  The investigators will use the patient satisfaction questionnaire within 10-15 days after discharge. The participants will be asked how useful the participants found the intervention, on a 0 to 10 scale, with 0 being not useful at all and 10 being extremely useful.

OTHER OUTCOMES:
30-day Hospital Readmissions | Discharge to 30 days after discharge
  The investigators will assess whether study participants had a hospital re-admission within 30 days of discharge using the Electronic Health Record

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer S Temel, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation